CLINICAL TRIAL: NCT02038543
Title: Influence of Hydroxyproline Plasma Concentration on Its Metabolism to Oxalate
Brief Title: Hydroxyproline Influence on Oxalate Metabolism
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Rare Diseases Clinical Research Network (Network); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, John Lieske, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-000150; U54DK083908 (NIH)
Record Dates: First submitted 2013-12-19; First posted 2014-01-16 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Hyperoxaluria
Keywords: Hyperoxaluria; Oxalate; Primary Hyperoxaluria
MeSH Terms: conditions — Hyperoxaluria; Hyperoxaluria, Primary | interventions — Hydroxyproline; Leucine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Primary hyperoxaluria patients (Experimental): Subjects will be infused with 13C5-hydroxyproline and 2H3-leucine for 6 hrs in the Clinical Research and Trials Unit (CRTU). The metabolic flux of 2H3-leucine has been well characterized, and is used as a control when studying the metabolism of trace infusions of labeled amino acids 3. Blood samples will be obtained every 30 min to determine the enrichment of plasma with 13C5-hydroxyproline and 2H3-leucine. Urine collections will be obtained hourly. The fluxes of whole body hydroxyproline and leucine will be calculated
  Interventions: Drug: Hydroxyproline and Leucine

INTERVENTIONS:
Drug: Hydroxyproline and Leucine — Subjects will be infused with 13C5-hydroxyproline and 2H3-leucine for 6 hrs in the CRTU. The metabolic flux of 2H3-leucine has been well characterized, and is used as a control when studying the metabolism of trace infusions of labeled amino acids 3. Blood samples will be obtained every 30 min to determine the enrichment of plasma with 13C5-hydroxyproline and 2H3-leucine. Urine collections will be obtained hourly. The fluxes of whole body hydroxyproline and leucine will be calculated
  Other Names: 13C5-hydroxyproline; 2H3-leucine

SUMMARY:
Primary hyperoxaluria is an inborn error of metabolism that results in marked overproduction of oxalate by the liver. The excess oxalate causes kidney failure and can cause severe systemic disease due to oxalate deposition in multiple body tissues.

Metabolic pathways that lead to oxalate are poorly understood, but recent evidence suggests that hydroxyproline may play a role. Sources of hydroxyproline include the diet and bone turnover. If hydroxyproline can be confirmed as a significant factor in primary hyperoxaluria, diet modification might be of value in reducing the severity of disease.

This protocol, in which hydroxyproline labelled with a cold isotope is infused intravenously in patients with primary hyperoxaluria, will allow the researchers to measure the amount of oxalate produced from hydroxyproline. The contribution of hydroxyproline metabolism to the amount of oxalate excreted in urine in will be able to be determined for patients with each of the known types of primary hyperoxaluria.

DETAILED DESCRIPTION:
The purpose of this study is to determine the contribution of hydroxyproline metabolism to urinary oxalate and glycolate excretion in patients with primary hyperoxaluria.

Oxalic acid (COOH)2 is an end product of metabolism that is synthesized mainly in the liver. The researchers have estimated that 10 - 20 mg is synthesized in the body of healthy adults each day. The main precursor of oxalate is glyoxylate (CHO•COOH). The bulk of the glyoxylate formed is normally transaminated to glycine (NH2•CH2•COOH) by alanine: glyoxylate aminotransferase (AGT) or reduced to glycolate (CHOH•COOH) by glyoxylate reductase (GR). Less than 10% of the glyoxylate is oxidized to oxalate by lactate dehydrogenase (LDH). In individuals with the disease, primary hyperoxaluria, AGT, GR, or hydroxy-oxoglutarate aldolase (HOGA) enzyme is deficient and the amount of oxalate synthesized by the liver increases to 80 - 300 mg per day. The increased oxalate excreted in urine can cause damage to kidney tissue. Calcium oxalate stones may form in the kidney or calcium oxalate crystals may deposit in renal tubules and the renal parenchyma (nephrocalcinosis). An increased rate of oxalate synthesis could also contribute to idiopathic calcium oxalate stone disease. Understanding the pathways of endogenous oxalate synthesis and identifying strategies that decrease oxalate production could be beneficial for individuals with these diseases.

Hydroxyproline is the primary source of glyoxylate identified in the body. Daily collagen turnover of bone results in the formation of 300 - 450 mg of hydroxyproline, which cannot be re-utilized by the body and is broken down. This metabolism yields 180 - 250 mg of glyoxylate. Further hydroxyproline is obtained from the diet, primarily from meat and gelatin-containing products. The bulk of the glyoxylate formed is converted to glycine by the liver enzyme AGT, some to glycolate and a small amount to oxalate. The proportion of these metabolites is not known with any certainty. In this study, a quantitative estimate of the metabolites formed will provide estimates of the contribution of hydroxyproline turnover to daily oxalate production.

ELIGIBILITY:
Inclusion criteria:

* Confirmed diagnosis of primary hyperoxaluria (PH)
* Estimated Glomerular Filtration Rate (eGFR) (by serum creatinine) > 50ml/min/1.73m^2 - Patients with a diagnosis of PH I, PH II, PH III, or Non I/Non II/Non III PH (PH types will be confirmed by DNA)

Exclusion criteria:

* eGFR < 50 ml/min/1.73m^2
* History of liver or kidney transplant
* Primary hyperoxaluria patients who have responded to pyridoxine therapy with reduction of urine oxalate excretion to < 0.45 mmol/1.73m^2/day
* Pregnancy

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-09; Primary Completion 2016-09 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Lieske, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Hyperoxaluria Center, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at Mayo Clinic in Rochester, Minnesota.
Groups:
- PH Type 1: In primary hyperoxaluria type 1, kidney stones typically begin to appear anytime from childhood to early adulthood, and end stage renal disease (ESRD) can develop at any age.
- PH Type 2: Primary hyperoxaluria type 2 is similar to type 1, but end stage renal disease (ESRD) develops later in life.
- PH Type 3: In primary hyperoxaluria type 3, affected individuals often develop kidney stones in early childhood, but few cases of this type have been described so additional signs and symptoms of this type are unclear.
- PH Type Non 1,2,3: Subjects who presented with overproduction of oxalate, leading to recurrent kidney and bladder stones, but are not identified as primary hyperoxaluria (PH) types 1, 2, or 3.
Period: Overall Study
Arm/Group | PH Type 1 | PH Type 2 | PH Type 3 | PH Type Non 1,2,3
Started | 7 | 4 | 8 | 3
Completed | 7 | 4 | 8 | 1
Not Completed | 0 | 0 | 0 | 2
Not completed — Screen Failure | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- PH Type Non 1,2,3: Subjects who presented with overproduction of oxalate, leading to recurrent kidney and bladder stones, but are not identified a PH types 1, 2, or 3.
- Total: Total of all reporting groups
Arm/Group | PH Type 1 | PH Type 2 | PH Type 3 | PH Type Non 1,2,3 | Total
Number analyzed (Participants) | 7 | 4 | 8 | 3 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 7 | 3 | 20
  >=65 years | 0 | 1 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 0 | 1 | 8
  Male | 4 | 0 | 8 | 2 | 14
Region of Enrollment [Number; unit: participants]
  United States | 7 | 4 | 8 | 3 | 22

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Conversion of Hydroxyproline (Hyp) to Urinary Oxalate (UOx)
Description: The overall contribution of hydroxyproline catabolism to urinary oxalate (UOx) and glycolate (UGlc) excretion is determined by the excess mole percent enrichment of urine with 13C2-oxalate and glycolate corrected for the fraction of labelled [15N,13C5]-Hyp that is circulating in the plasma.
Time Frame: Participants will be followed for the duration of study infusion and observation, an average of 24 hours.
Population: 2 subjects from the PH Type Non 1,2,3 withdrew from the study. Subjects with PH Type Non 1,2,3 were not included in the analysis as only 1 subject completed the study.
Measure: Mean (Standard Error); unit: percent converted
Groups:
- PH Type Non 1,2,3: Subjects who presented with overproduction of oxalate, leading to recurrent kidney and bladder stones, but are not identified as PH types 1, 2, or 3.
Arm/Group | PH Type 1 | PH Type 2 | PH Type 3 | PH Type Non 1,2,3
Number analyzed (Participants) | 7 | 4 | 8 | 0
percent converted | 12.8 (4.7) | 32.9 (8.0) | 14.8 (1.8) |

2. Secondary Outcome: Mean Percent Conversion of Hydroxyproline (Hyp) to Urinary Glycolate (UGIc)
Description: The overall contribution of Hyp catabolism to urinary oxalate (UOx) and glycolate (UGlc) excretion is determined by the excess mole percent enrichment of urine with 13C2-oxalate and glycolate corrected for the fraction of labelled [15N,13C5]-Hyp that is circulating in the plasma.
Time Frame: Participants will be followed for the duration of the study infusion and observations, an average of 24 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percent converted
Arm/Group | PH Type 1 | PH Type 2 | PH Type 3 | PH Type Non 1,2,3
Number analyzed (Participants) | 7 | 4 | 8 | 0
percent converted | 16.3 (4.0) | 1.4 (0.4) | 2.5 (1.3) |

ADVERSE EVENTS:
Time Frame: Participants were followed for the duration of study infusion and observation, an average of 24 hours.
Arm/Group | PH Type 1 | PH Type 2 | PH Type 3 | PH Type Non 1,2,3
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/4 | 0/8 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/4 | 0/8 | 0/1
Other Adverse Events (participants affected / at risk) | 0/7 | 0/4 | 0/8 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes